CLINICAL TRIAL: NCT03113617
Title: 68Ga-RM2 PET/CT for Detection of Regional Nodal and Distant Metastases in Patients With Intermediate and High-Risk Prostate Cancer
Brief Title: 68Ga-RM2 PET/CT in Detecting Regional Nodal and Distant Metastases in Patients With Intermediate or High-Risk Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andrei Iagaru (Other)
Responsible Party: Sponsor-Investigator, Andrei Iagaru, Associate Professor of Radiology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-40373; NCI-2017-00547 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PROS0077 (Other: OnCore); IRB-40373 (Other: Stanford IRB)
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Results first posted 2023-05-24 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Stage II Prostate Adenocarcinoma; Stage III Prostate Adenocarcinoma; Stage IV Prostate Adenocarcinoma
MeSH Terms: interventions — BAY 86-7548; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (68Ga-RM2 PET/CT) (Experimental): Patients receive 68Ga-RM2 IV. Within 45-60 minutes, patients undergo a PET/CT scan. Patients may undergo a second PET/CT scan immediately after the first scan for attenuation correction. Patients may undergo also a repeat 68Ga-RM2 PET/CT scan after the completion of their treatment to evaluate response to therapy, if requested by the treating physician.
  Interventions: Procedure: Computed Tomography; Drug: Gallium Ga 68-labeled GRPR Antagonist BAY86-7548; Other: Laboratory Biomarker Analysis; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT SCAN; tomography
Drug: Gallium Ga 68-labeled GRPR Antagonist BAY86-7548 — Given IV
  Other Names: (68)Ga-DOTA-4-amino-1-carboxymethylpiperidine-d-Phe-Gln-Trp-Ala-Val-Gly-His-Sta-Leu-NH2; 68Ga-Bombesin Antagonist BAY86-7548; 68Ga-DOTA RM2; 68Ga-DOTA-Bombesin Analog BAY86-7548; [68Ga]-labeled Bombesin Analog BAY86-7548; [68Ga]RM2; BAY 86-7548; Ga-68-labeled Bombesin Antagonist BAY 86-7548; Gallium Ga68-labeled GRPR Antagonist RM2
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase II trial studies how well gallium Ga 68-labeled gastrin-releasing peptide receptor (GRPR) antagonist BAY86-7548 (68Ga-RM2) positron emission tomography (PET)/computed tomography (CT) works in detecting regional nodal and distant metastases in patients with intermediate or high-risk prostate cancer. 68Ga-RM2 PET/CT scan may be able to see smaller tumors than the standard of care CT or magnetic resonance imaging scan.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate 68Ga-RM2 PET/CT for detection of intermediate and high-risk prostate cancer prior to prostatectomy.

OUTLINE:

Patients receive 68Ga-RM2 intravenously (IV). Within 45-60 minutes, patients undergo a PET/CT scan. Patients may undergo a second PET/CT scan immediately after the first scan for attenuation correction. Patients may undergo also a repeat 68Ga-RM2 PET/CT scan after the completion of their treatment to evaluate response to therapy, if requested by the treating physician.

After completion of study, patients are followed up at 24-48 hours and within 3-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven prostate adenocarcinoma
* Planned prostatectomy with lymph node dissection
* Intermediate to high-risk disease (as determined by elevated PSA [PSA > 10], T-stage [T2b or greater], Gleason score [Gleason score > 6] or other risk factors)
* Able to provide written consent
* Karnofsky performance status of >= 50 (or Eastern Cooperative Oncology Group [ECOG]/World Health Organization [WHO] equivalent)
* Diagnostic CT or magnetic resonance imaging (MRI) performed within 30 days prior to the 68Ga-RM2 PET

Exclusion Criteria:

* Inability to lie still for the entire imaging time (approximately 30 minutes)
* Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.)
* Any additional medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2021-12-19 (Actual); Study Completion 2021-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Iagaru, Principal Investigator — Stanford Cancer Institute
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duan H, Davidzon GA, Moradi F, Liang T, Song H, Iagaru A. Modified PROMISE criteria for standardized interpretation of gastrin-releasing peptide receptor (GRPR)-targeted PET. Eur J Nucl Med Mol Imaging. 2023 Nov;50(13):4087-4095. doi: 10.1007/s00259-023-06385-z. Epub 2023 Aug 9. PMID 37555901

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (68Ga-RM2 PET/CT)
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (68Ga-RM2 PET/CT)
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 20
Age, Continuous [Mean (Standard Deviation); unit: participant] | 63 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 31
  More than one race | 1
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity, Specificity, Positive, and Negative Predictive Value of 68Ga-RM2 PET for the Detection of Regional Nodal Metastases Compared to Pathology at Radical Prostatectomy
Description: True positive patient is defined as PET positive for regional nodes, pathology at prostatectomy positive for regional nodes or PET positive for regional nodes, pathology negative for regional nodes, imaging after prostatectomy demonstrates node was not removed at surgery, and follow-up biopsy or imaging demonstrates presence of nodal disease. True negative patient is defined as PET negative for regional nodes, pathology at prostatectomy negative for regional nodes. False positive patient is defined as PET positive for regional nodes, pathology at prostatectomy is negative, and imaging after prostatectomy
Time Frame: week 1 study visit following radiopharmaceutical administration, up to 2 hours to assess
Measure: Number (95% Confidence Interval); unit: percentage of cases
Arm/Group | Diagnostic (68Ga-RM2 PET/CT)
Number analyzed (Participants) | 44
percentage of cases
  Specificity | 55.6 [21.2 to 86.3]
  Sensitivity | 92.3 [74.9 to 99.1]
  Positive predictive value | 71.4 [29.0 to 96.3]
  Negative predictive value | 85.7 [67.3 to 96.0]

2. Secondary Outcome: Sensitivity, Specificity, Negative and Positive Predictive Value for Detection of Regional Nodal Metastases in Comparison to Cross Sectional Imaging Performed Contemporaneously With the 68Ga-RM2 PET
Description: as for outcome 1
Time Frame: week 1 study visit following radiopharmaceutical administration, up to 2 hours to assess
Measure: Number (95% Confidence Interval); unit: percentage of cases
Arm/Group | Diagnostic (68Ga-RM2 PET/CT)
Number analyzed (Participants) | 44
percentage of cases
  Sensitivity | 22.2 [2.8 to 60.0]
  Specificity | 96.2 [80.0 to 99.9]
  Positive predictive value | 66.7 [9.4 to 99.2]
  Negative predictive value | 78.1 [60.0 to 90.7]

3. Other Pre Specified Outcome: Incidence of Osseous and Distant Metastatic Lesions
Time Frame: Up to 3 years
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Maximum Standardized Uptake Value (SUVmax) From 68Ga-RM2 PET
Description: Correlation between SUVmax from gallium Ga 68-labeled GRPR antagonist BAY86-7548 PET and short axis diameter of nodal disease on cross sectional imaging correlate to presence of true pathology will be performed.
Time Frame: Up to 3 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: PSA Progression Free Survival
Description: Patients with and without pelvic nodal metastases will be compared.
Time Frame: At 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | Diagnostic (68Ga-RM2 PET/CT)
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT03113617/Prot_SAP_002.pdf